CLINICAL TRIAL: NCT06660368
Title: A Prospective, Multicenter, Randomized, Open-Label, Phase II Study of Salvage BCL2i Plus CLAG-M in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: BCL2i CLAG-M in R/R Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23154
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — Cladribine; Cytarabine; Mitoxantrone; Granulocyte Colony-Stimulating Factor; Clinical Protocols; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLAG-based therapy with venetoclax (Experimental): Study participants will receive CLAG-M (cladribine, cytarabine, G-CSF, mitoxantrone) and Venetoclax
  Interventions: Drug: Cladribine, Cytarabine, Mitoxantrone, G-CSF (CLAG-M) regimen; Drug: Venetoclax
- CLAG-based therapy without venetoclax (Active Comparator): Study participants will receive CLAG-M (cladribine, cytarabine, G-CSF, mitoxantrone)
  Interventions: Drug: Cladribine, Cytarabine, Mitoxantrone, G-CSF (CLAG-M) regimen

INTERVENTIONS:
Drug: Cladribine, Cytarabine, Mitoxantrone, G-CSF (CLAG-M) regimen — Filgrastim/G-CSF 300 mcg/day for 6 days beginning 24 hours prior to multiagent chemotherapy (days 0-5), cladribine 5 mg/m2 given intravenously over 2 hours for 5 consecutive days (days 1-5), cytarabine given IV over 4 hours for 5 consecutive days (days 1-5) beginning 2 hours after the completion of cladribine, and mitoxantrone 16 mg/m2 given intravenously over 30 minutes for 3 days (days 1-3) after completion of cytarabine.
Drug: Venetoclax — Venetoclax will be administered orally, once daily, with food.
  Arms: CLAG-based therapy with venetoclax

SUMMARY:
This multicenter, open-label phase II study combines CLAG-based therapy with or without venetoclax in patients with relapsed or refractory (R/R) acute myeloid leukemia (AML) in order to improve measurable residual disease (MRD) clearance and event-free survival. Investigators hypothesize that the addition of venetoclax to CLAG-M in patients with relapsed or refractory AML is safe, and superior to CLAG-M alone in improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Ability to understand and stated willingness to comply with all study procedures and availability for the duration of the study.
* Adults aged ≥18 years - 80 years.
* Patients with documented refractory or relapsed AML: Refractory disease is defined as failure to achieve CR (i.e., <5% blasts in BM or blood) with or without normal restoration of hematopoiesis (Cri) after at least 1 cycle of intensive induction therapy (or 2 cycles of non-intensive induction). Relapse: Recurrence of disease after achieving remission, meeting one or more of the following criteria: ≥ 5% blasts in the marrow or peripheral blood, extramedullary disease.
* Secondary AML arising out of MDS previously treated with HMA, HMA + venetoclax (if > 3 months from venetoclax exposure), and/or 1 cycle of induction chemotherapy.
* Extramedullary AML with marrow involvement is allowed as long as concurrent medullary AML is present.
* ECOG performance status ≤ 2.
* Participants must have adequate organ function as defined within the protocol.
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Testing is not mandatory.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and have an undetectable HCV viral load. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. Testing is not mandatory.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 4 months after completion of study drug administration.

Exclusion Criteria:

* Venetoclax-refractory disease or recent venetoclax exposure < 3 months prior to first dose of study therapy.
* Prior treatment with a high-dose cytarabine-containing regimen (e.g., no prior CLAG/FLAG/MEC/CLIA/HAM, etc.).
* Allogeneic stem cell transplant in the past 3 months.
* Less than 14 days from last AML-directed therapy or five half-lives, whichever is shorter, not including hydroxyurea.
* Known history of prior TP53 mutation (results from any myeloid mutation panel are not required for screening eligibility).
* Active CNS involvement by AML.
* WBC count ≥25k at the time study treatment begins.
* Uncontrolled intercurrent systemic illness that would limit compliance.
* Concurrent malignancy in addition to AML that requires active treatment with some exceptions.
* Immunosuppressive therapy in the past 14 days except for prednisone at ≤ 10 mg/day or equivalent AND no active or uncontrolled graft-versus-host disease (GvHD).
* Participants who have not recovered from adverse events (Aes) due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1), with the exception of alopecia.
* Participants who are receiving any other investigational agents.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with active heart disease that limits the use of mitoxantrone or recent (<6 months) history of an acute cardiovascular event (STEMI, NSTEMI).
* Pregnant women are excluded from this study because venetoclax, cladribine, and cytarabine are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these drugs, breastfeeding should be discontinued.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
MRD-Negative Remission Rate | Up to 18 months
  The rate of MRD negative remission will be calculated for each arm.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 18 months
  EFS will be measured from the date of randomization to the first of:
  failure to achieve composite CR by the end of induction, relapse after achieving composite CR, or death from any cause
Treatment-Related Toxicities | Up to 18 months
  The number of participants who experience an AE or SAE.
Overall survival (OS) based on treatment arm | Up to 18 months
  OS is defined as time from treatment initiation to death or last follow-up if alive at last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: David Sallman, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts